CLINICAL TRIAL: NCT01453933
Title: Phase IV, Randomized, Open Label, Crossover, Intervention Trial to Investigate the Effect of the Switch of Lopinavir/Ritonavir to Raltegravir on Endothelial Function, Chronic Inflammation, Immune Activation and HIV Replication <50 Copies/ml
Brief Title: RAltegravir Switch STudy: Effects on Endothelial Recovery
Acronym: RASSTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, S.F.L. van Lelyveld, principal investigator, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RASSTER2010
Record Dates: First submitted 2011-10-10; First posted 2011-10-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infection; Endothelial Dysfunction
Keywords: Anti-HIV Agents; Anti-Retroviral Agents; Antiviral Agents; Anti-Infective Agents; Lopinavir/ritonavir
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltegravir (Active Comparator): At baseline, lopinavir-ritonavir will be switched to raltegravir (cross-over after 8 weeks).
  Interventions: Drug: raltegravir
- Lopinavir/ritonavir (No Intervention): Subjects will continue lopinavir/ritonavir (cross-over after 8 weeks)

INTERVENTIONS:
Drug: raltegravir — Switch of lopinavir/ritonavir to raltegravir 400 mg BID (duration 8 weeks)
  Other Names: Isentress
  Arms: Raltegravir

SUMMARY:
Treatment with HIV-infection with protease inhibitors is associated with high blood lipids and higher chance for cardiovascular complications. The RASSTER study aims to investigate the effect of switching the protease inhibitor lopinavir/ritonavir to raltegravir on vessel wall function and inflammation,and activation of the immune system. we hypothesize that with this intervention these parameters will improve. Since decreased vessel wall function and inflammation are initial steps in the process of atherosclerosis, it is important to know this data when treating HIV-infected patients.

DETAILED DESCRIPTION:
Fixed dose combination lopinavir/ritonavir (LPV/r) is a widespread used antiretroviral drug belonging to the class of protease inhibitors (PIs). PIs are associated with an increased risk of myocardial infarction. However, data is available suggesting increased levels of plasma lipids are not the sole explanation for this observation. Treatment with LPV/r might lead to a decrease of endothelial function as well, thus explaining the increased risk of myocardial infarction besides increased plasma lipids. Raltegravir is a registered antiretroviral drug with no known cardiovascular side effects. We hypothesize that switching LPV/r to raltegravir in HIV-infected patients with suppressed plasma viral load (<50 copies/ml) will lead to an improvement of endothelial function.

Objective:

* First, to assess the effect of the switch of lopinavir/ritonavir to raltegravir on endothelial function.
* Second, to assess the effect of the intervention mentioned above on markers of endothelial function; immune activation; chronic inflammation; and, on plasma HIV-RNA below the cut-off of 50 copies/ml.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* HIV-1 infection
* Treatment with antiretroviral regimen containing lopinavir/ritonavir for at least the previous 3 months
* No other protease inhibitors besides lopinavir/ritonavir in antiretroviral regimen
* Subjects must have a minimum period of viral suppression (plasma HIV-RNA < 50 copies/ml) of 6 months
* Subjects will not have a history of virological failure on antiretroviral therapy
* Results of previous resistance testing allowing replacement of lopinavir/ritonavir by raltegravir
* CD4+ cell count > 200 cells/µL
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Raltegravir hypersensitivity
* Treatment of underlying malignancy
* Renal insufficiency requiring dialysis
* Acute or decompensated chronic hepatitis (Child-Pugh score C)
* Modification of antiretroviral regimen in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in flow mediated dilatation (FMD) of the brachial artery | week 8, week16
  Change in flow-mediated dilatation (FMD) of the brachial artery after 8 weeks of raltegravir treatment as compared to the control group (treatment with lopinavir/ritonavir)

SECONDARY OUTCOMES:
Change in markers of chronic inflammation | Baseline, week 2, week 4, week 8, week 10, week 12 and week 16
Change in markers of immune activation | Baseline, week 2, week 4, week 8, week 10, week 12 and week 16
Change in markers of endothelial function | Baseline, week 2, week 4, week 8, week 10, week 12 and week 16
Changes in plasma HIV-RNA below 50 copies/ml | Baseline, week 8, week 16

CONTACTS AND LOCATIONS:
Overall Officials: Andy IM Hoepelman, MD, Principal Investigator — University Medical Center Utrecht, The Netherlands; Steven FL van Lelyveld, MD, Study Director — University Medical Center Utrecht, The Netherlands
Locations (2):
- Netherlands (2):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Krikke M, Tesselaar K, van den Berk GEL, Otto SA, Freriks LH, van Lelyveld SFL, Visseren FJL, Hoepelman AIM, Arends JE. The effect of switching protease inhibitors to raltegravir on endothelial function, in HIV-infected patients. HIV Clin Trials. 2018 Apr;19(2):75-83. doi: 10.1080/15284336.2018.1455366. PMID 29770748